CLINICAL TRIAL: NCT01161628
Title: Phase II Trial Evaluating the Safety and Efficacy of Rituximab as Primary Treatment for Extensive Chronic Graft Versus Host Disease
Brief Title: Rituximab for the Primary Treatment of Denovo Extensive Chronic Graft Versus Host Disease (GVHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Blood and Marrow Transplant Group of Georgia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 893
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: Chronic Graft versus Host Disease; allogeneic stem cell transplant
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituxan (Experimental): All patients receive Rituximab 375 mg/m2/dose x 4 weekly doses on days 1, 8, 15 and 22 and then at 3, 6, 9 and 12 months.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2/dose x 4 weekly doses on days 1, 8, 15 and 22 and then at 3, 6, 9 and 12 months.
  Other Names: Rituxan

SUMMARY:
Rituximab is an attractive agent to bring to the upfront treatment of chronic graft-versus-host disease (cGVHD) due to its favorable toxicity profile, its proven efficacy in the treatment of steroid-refractory cGVHD, and its ability to serve as a steroid sparing agent in other autoimmune diseases. The investigators hope to demonstrate that Rituximab has significant activity in cGVHD when utilized early in the course of the process. In addition, the investigators hope to show that the early use of Rituximab may allow for the earlier discontinuation of immunosuppression while obviating the need for long courses of systemic corticosteroids, which should translate into reduced treatment-related morbidity and mortality associated with cGVHD.

DETAILED DESCRIPTION:
Although allogeneic hematopoietic stem cell transplantation (HSCT) remains an important curative therapy for many patients with hematological malignancies, treatment-related morbidity and mortality continue to be a major challenge. Chronic GVHD remains a major complication following allogeneic HSCT, with more than half of patients being affected. Although cGVHD has been associated with decreased relapse risk due to the well documented graft-versus-malignancy effect, it is also associated with significant adverse consequences in terms of morbidity, mortality, quality-of-life, and treatment costs associated with HSCT.

Rituximab has been investigated in a small number of patients with refractory cGVHD using the standard regimen of 375 mg/m2/week for 4 weeks. Ratanatharathorn et al. documented a sustained response in four of eight patients with steroid-refractory cGVHD with diffuse or localized sclerodermatous manifestations. Similarly, Canninga-vanDijk et al. and Okamoto et al. observed cases with clinical, laboratory and histological improvement after Rituximab treatment. Cutler et al. reported the results of their phase I-II study with Rituximab in 21 patients with steroid-refractory cGVHD. Treatment was well tolerated, and toxicity limited to infectious events, without any hematological toxicities and only a significant reduction in circulating immunoglobulins documented after therapy. Objective responses were documented in 70% of patients (including 10% complete response) primarily for those with skin and musculoskeletal involvement, allowing tapering, and in some cases withdrawing, of previous immunosuppressant therapy. A correlation between clinical response and decrease in the titre of antibodies against Y chromosome-encoded minor HLA antigens was shown. The results of these preliminary studies highlight the potential therapeutic activity of Rituximab on some cGVHD manifestations and a particularly high efficacy for skin involvement, including scleroderma. Recently, Zaja et al. confirmed the activity of Rituximab in refractory cGVHD in a larger series of 38 patients. Treatment was generally well tolerated and nearly 60% and 50% of patients had a clinical improvement of their skin and mouth manifestations, respectively. The median time-to-response was nearly 2 months and in some cases responses were durable. Responses were also detectable in some patients with eye, liver, lung, gut and joint involvement, allowing reduction and/or suspension of previous baseline immunosuppressive therapy in a significant number of patients

ELIGIBILITY:
Inclusion Criteria:

* First episode of extensive chronic GvHD, without residual or concurrent acute GvHD.
* Age 18 - 75
* Any primary diagnosis requiring treatment by allogeneic HSCT
* Recipient of an allogeneic stem cell transplant (bone marrow, peripheral blood stem cell, or cord blood) from a related or unrelated donor, minimum 80 days ago
* Conditioning regimen: Myeloablative or non-myeloablative
* Patient gives written informed consent

Exclusion Criteria:

* Creatinine > 2.0 mg/dl
* Uncontrolled, active infection
* Recurrent or progressive malignancy
* Anticipated life expectancy of less than 1 year
* Pregnant or breast feeding
* Contraindications to administration of the study intervention or known inability of the patient to tolerate the study intervention
* Patients with perceived fixed, irreversible defects (pulmonary involvement, contractures, etc.) which would not be expected to improve with the study intervention
* Residual or concurrent acute GVHD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2014-01 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Solomon, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canninga-van Dijk MR, van der Straaten HM, Fijnheer R, Sanders CJ, van den Tweel JG, Verdonck LF. Anti-CD20 monoclonal antibody treatment in 6 patients with therapy-refractory chronic graft-versus-host disease. Blood. 2004 Oct 15;104(8):2603-6. doi: 10.1182/blood-2004-05-1855. Epub 2004 Jul 13. PMID 15251978
- [Background] Ratanatharathorn V, Carson E, Reynolds C, Ayash LJ, Levine J, Yanik G, Silver SM, Ferrara JL, Uberti JP. Anti-CD20 chimeric monoclonal antibody treatment of refractory immune-mediated thrombocytopenia in a patient with chronic graft-versus-host disease. Ann Intern Med. 2000 Aug 15;133(4):275-9. doi: 10.7326/0003-4819-133-4-200008150-00011. PMID 10929168
- [Background] Ratanatharathorn V, Ayash L, Reynolds C, Silver S, Reddy P, Becker M, Ferrara JL, Uberti JP. Treatment of chronic graft-versus-host disease with anti-CD20 chimeric monoclonal antibody. Biol Blood Marrow Transplant. 2003 Aug;9(8):505-11. doi: 10.1016/s1083-8791(03)00216-7. PMID 12931119
- [Background] Okamoto M, Okano A, Akamatsu S, Ashihara E, Inaba T, Takenaka H, Katoh N, Kishimoto S, Shimazaki C. Rituximab is effective for steroid-refractory sclerodermatous chronic graft-versus-host disease. Leukemia. 2006 Jan;20(1):172-3. doi: 10.1038/sj.leu.2403996. No abstract available. PMID 16239908
- [Background] Zaja F, Bacigalupo A, Patriarca F, Stanzani M, Van Lint MT, Fili C, Scime R, Milone G, Falda M, Vener C, Laszlo D, Alessandrino PE, Narni F, Sica S, Olivieri A, Sperotto A, Bosi A, Bonifazi F, Fanin R; GITMO (Gruppo Italiano Trapianto Midollo Osseo). Treatment of refractory chronic GVHD with rituximab: a GITMO study. Bone Marrow Transplant. 2007 Aug;40(3):273-7. doi: 10.1038/sj.bmt.1705725. Epub 2007 Jun 4. PMID 17549053
- [Background] Cutler C, Miklos D, Kim HT, Treister N, Woo SB, Bienfang D, Klickstein LB, Levin J, Miller K, Reynolds C, Macdonell R, Pasek M, Lee SJ, Ho V, Soiffer R, Antin JH, Ritz J, Alyea E. Rituximab for steroid-refractory chronic graft-versus-host disease. Blood. 2006 Jul 15;108(2):756-62. doi: 10.1182/blood-2006-01-0233. Epub 2006 Mar 21. PMID 16551963
- [Background] Stewart BL, Storer B, Storek J, Deeg HJ, Storb R, Hansen JA, Appelbaum FR, Carpenter PA, Sanders JE, Kiem HP, Nash RA, Petersdorf EW, Moravec C, Morton AJ, Anasetti C, Flowers ME, Martin PJ. Duration of immunosuppressive treatment for chronic graft-versus-host disease. Blood. 2004 Dec 1;104(12):3501-6. doi: 10.1182/blood-2004-01-0200. Epub 2004 Aug 3. PMID 15292060
- [Background] Lee SJ, Vogelsang G, Flowers ME. Chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2003 Apr;9(4):215-33. doi: 10.1053/bbmt.2003.50026. PMID 12720215

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituxan: all patients will receive Rituxan for the treatment of newly diagnosed chronic GVHD
  Rituximab: Rituximab 375 mg/m2/dose x 4 weekly doses on days 1, 8, 15 and 22 and then at 3, 6, 9 and 12 months.
Period: Overall Study
Arm/Group | Rituxan
Started | 25
Completed | 17
Not Completed | 8
Not completed — Death | 6
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rituxan
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Race/Ethnicity, Customized [Number; unit: participants]
  White | 21
  Black/African American | 4

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Response of cGVHD to Treatment.
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Rituxan
Number analyzed (Participants) | 22
percentage of patients | 84
Statistical Analysis 1: Comparison: Rituxan; Null hypothesis: p (CR rate) is 0.5 or less versus... Alternative hypothesis: p >0.5 A sample size of 25 patients gives 90% power with an alpha = 0.05; Test type: Superiority or Other; p < 0.5, t-test, 2 sided

2. Secondary Outcome: Requirement for Systemic Corticosteroid Use
Time Frame: 2 years
Population: 20 out of the 25 patients enrolled received no corticosteroids at all during the course of treatment for cGVHD
Measure: Number; unit: participants
Arm/Group | Rituxan
Number analyzed (Participants) | 25
participants | 20

3. Secondary Outcome: Time to Immunosuppression Withdrawal
Time Frame: 2 years
Measure: Median (Full Range); unit: days
Arm/Group | Rituxan
Number analyzed (Participants) | 17
days | 300 [138 to 488]

4. Secondary Outcome: Incidence of Overall Survival
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Rituxan
Number analyzed (Participants) | 25
percentage of patients | 82

5. Primary Outcome: Rate of Overall Response of cGVHD to Treatment
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Rituxan
Number analyzed (Participants) | 22
percentage of patients | 88

6. Primary Outcome: Rate of Partial Response of cGVHD to Treatment
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Rituxan
Number analyzed (Participants) | 22
percentage of patients | 5

7. Secondary Outcome: Duration of Systemic Corticosteroid Use
Time Frame: 2 years
Population: Only 2 patients out of the 22 evaluable patients enrolled received steroids during the course of treatment for cGVHD. A total of 25 patients were enrolled; 3 patients were excluded from this analysis due to treatment failure.
Measure: Median (Full Range); unit: days
Arm/Group | Rituxan
Number analyzed (Participants) | 2
days | 15 [13 to 18]

8. Secondary Outcome: Incidence of Disease-free Survival
Time Frame: 2 years
Population: Of the surviving patients at 2 years (82% of initial enrolled population)
Measure: Number; unit: percentage of patients
Arm/Group | Rituxan
Number analyzed (Participants) | 20
percentage of patients | 79

9. Secondary Outcome: Incidence of Non-relapse Mortality
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Rituxan
Number analyzed (Participants) | 25
percentage of patients | 21

ADVERSE EVENTS:
Time Frame: adverse event data was collected for 2 years.
Arm/Group | Rituxan
Serious Adverse Events (participants affected / at risk) | 17/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituxan (N=25)
Failure to thrive (General disorders) | 1 (1)
Ischemic cardiomyopathy (Cardiac disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Liver dysfunction (Hepatobiliary disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
altered mental status (Psychiatric disorders) | 1 (1)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Fever (Investigations) | 13 (13)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituxan (N=25)
abdominal discomfort (Gastrointestinal disorders) | 4
abdominal distention (Gastrointestinal disorders) | 3
abdominal pain (Gastrointestinal disorders) | 6
muscle aches (Musculoskeletal and connective tissue disorders) | 3
acute renal failure (Renal and urinary disorders) | 3
hypoalbuminemia (Hepatobiliary disorders) | 6
increased alkaline phosphatase (Hepatobiliary disorders) | 5
increased ALT (Hepatobiliary disorders) | 10
altered mental status (Nervous system disorders) | 3
neutropenia (Blood and lymphatic system disorders) | 20
anemia (Blood and lymphatic system disorders) | 14
anorexia (Gastrointestinal disorders) | 13
anxiety (Psychiatric disorders) | 4
increased AST (Hepatobiliary disorders) | 10
back pain (Musculoskeletal and connective tissue disorders) | 5
shoulder pain (Musculoskeletal and connective tissue disorders) | 3
bacteremia (Infections and infestations) | 2
BKV cystitis (Renal and urinary disorders) | 2
blurry vision (Eye disorders) | 2
bruising (Blood and lymphatic system disorders) | 2
cardiomyopathy (Cardiac disorders) | 3
chest congestion (Respiratory, thoracic and mediastinal disorders) | 3
chest pain (Cardiac disorders) | 4
chills (Investigations) | 2
conjunctivitis (Eye disorders) | 3
constipation (Gastrointestinal disorders) | 2
cough (Respiratory, thoracic and mediastinal disorders) | 11
crackles at lung bases (Respiratory, thoracic and mediastinal disorders) | 2
hypercreatinemia (Renal and urinary disorders) | 2
deconditioned (Investigations) | 6
dehydration (Endocrine disorders) | 2
depression (Psychiatric disorders) | 5
diarrhea (Gastrointestinal disorders) | 13
diminished breath sounds (Respiratory, thoracic and mediastinal disorders) | 3
dizziness (Nervous system disorders) | 2
drowsiness (Nervous system disorders) | 2
dry eyes (Eye disorders) | 4
dry lips (Investigations) | 3
dry mouth (Gastrointestinal disorders) | 10
dry skin (Skin and subcutaneous tissue disorders) | 4
dysuria (Renal and urinary disorders) | 7
ear pain (Ear and labyrinth disorders) | 2
edema (Cardiac disorders) | 8
buccal mucosa erythema (Gastrointestinal disorders) | 3
erythematous lesion (Skin and subcutaneous tissue disorders) | 2
extremity pain (Musculoskeletal and connective tissue disorders) | 3
eye drainage (Eye disorders) | 3
eye irritation (Eye disorders) | 3
fatigue (Investigations) | 17
fever (Investigations) | 6
food intolerance (Gastrointestinal disorders) | 3
gastritis (Gastrointestinal disorders) | 3
GVHD - gut (Gastrointestinal disorders) | 3
GVHD - oral (Gastrointestinal disorders) | 5
GVHD - skin (Skin and subcutaneous tissue disorders) | 2
hematuria (Renal and urinary disorders) | 4
hemorrhoids (Gastrointestinal disorders) | 2
hypercalcemia (Metabolism and nutrition disorders) | 2
hyperglycemia (Metabolism and nutrition disorders) | 13
hyperkalemia (Metabolism and nutrition disorders) | 8
hypernatremia (Metabolism and nutrition disorders) | 3
hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
hypertension (Cardiac disorders) | 6
hypocalcemia (Metabolism and nutrition disorders) | 6
hypokalemia (Metabolism and nutrition disorders) | 7
hypomagnesemia (Metabolism and nutrition disorders) | 2
hyponatremia (Metabolism and nutrition disorders) | 4
hypotension (Cardiac disorders) | 3
hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
insomnia (Nervous system disorders) | 6
joint pain (Musculoskeletal and connective tissue disorders) | 4
joint stiffness (Musculoskeletal and connective tissue disorders) | 4
lethargy (Investigations) | 5
lichenoid changes in mouth (Gastrointestinal disorders) | 5
lip lesion (Investigations) | 2
loss of coordination (Nervous system disorders) | 10
lower extremity edema (Cardiac disorders) | 2
lymphopenia (Blood and lymphatic system disorders) | 3
mastoiditis (Ear and labyrinth disorders) | 2
mouth pain (Gastrointestinal disorders) | 6
mouth sensitivity (Gastrointestinal disorders) | 10
mouth sores (Gastrointestinal disorders) | 2
mucositis (Gastrointestinal disorders) | 2
muscle pain (Musculoskeletal and connective tissue disorders) | 3
myalgia (Musculoskeletal and connective tissue disorders) | 2
nausea (Gastrointestinal disorders) | 10
oral lesions (Gastrointestinal disorders) | 2
catheter site pain (Investigations) | 2
parainfluenza (Infections and infestations) | 3
pelvic pain (Musculoskeletal and connective tissue disorders) | 2
peripheral neuropathy (Nervous system disorders) | 4
pleural effusions (Respiratory, thoracic and mediastinal disorders) | 2
pneumonia (Infections and infestations) | 4
pneumonitis (Infections and infestations) | 2
pruritus (Investigations) | 10
pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3
respiratory syncytial virus (Infections and infestations) | 3
rash (Skin and subcutaneous tissue disorders) | 11
rectal pain (Gastrointestinal disorders) | 2
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 2
rhinovirus (Infections and infestations) | 5
rhonchi (Respiratory, thoracic and mediastinal disorders) | 3
sepsis (Investigations) | 2
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 9
sinus congestion (Investigations) | 5
skin lesion (Skin and subcutaneous tissue disorders) | 3
sore throat (Gastrointestinal disorders) | 2
staph epi bacteremia (Infections and infestations) | 2
steroid-induced diabetes (Metabolism and nutrition disorders) | 2
stool urgency (Gastrointestinal disorders) | 3
tachycardia (Cardiac disorders) | 3
thrombocytopenia (Blood and lymphatic system disorders) | 9
tremors (Nervous system disorders) | 2
upper respiratory infection (Infections and infestations) | 3
urinary frequency (Renal and urinary disorders) | 2
urinary incontinence (Renal and urinary disorders) | 3
urinary tract infection (Infections and infestations) | 4
urinary urgency (Renal and urinary disorders) | 2
vaginal irritation (Reproductive system and breast disorders) | 2
vomiting (Gastrointestinal disorders) | 8
leukopenia (Blood and lymphatic system disorders) | 13
weakness (Investigations) | 13
weight loss (Metabolism and nutrition disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less